CLINICAL TRIAL: NCT00285883
Title: Directly Observed Therapy in High Risk Populations in Newark, NJ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Saint Michael's Medical Center (Other)
Collaborators: Hoffmann-La Roche (Industry)
Other Study IDs: 36/03
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2006-02-28 (Estimated); Status verified 2006-01

CONDITIONS: Directly Observed Therapy; HIV Infections
Keywords: Invirase; HIV; DOT; Treatment Experienced
MeSH Terms: conditions — Directly Observed Therapy; HIV Infections | interventions — Saquinavir; Ritonavir

INTERVENTIONS:
Drug: Invirase
Drug: Norvir

SUMMARY:
30 patients with poor antiretroviral therapy compliance will be identified from our pool of patients at Saint Michael's Medical Center and be given Directly observed therapy.

DETAILED DESCRIPTION:
30 patients with poor antiretroviral therapy compliance will be identified from our pool of patients at Saint Michael's Medical Center. Consent will be obtained, their regimens will be switched to QD based on previous therapies and resistance patterns if available. Patients will be placed on direct observed therapy.Each patient will be placed on Fortovase/Ritonavir (1600mg/100mg)QD plus two or three NRTIs based on a phenotypic baseline testing to a protease inhibitor. Patients will visit the office at baseline, weeks 1, 4, 8, 12, 16, 24, 32, 40, and 48. Patients will also be visited daily by the social worker (or designee) to observe patients taking their antiretroviral therapy for 6 months. After six months of direct observed therapy patients will be given a diary card to record administration of medications and the social worker ( or designee) will visit the home twice weekly. If the patient experiences a change in therapy secondary to virologic failure, the patient will return to baseline visit for the new once a day regimen. Virologic failure will be defined as < .5 log drop between each visit or > 400 copies/mL at week 24 on two separate occasions at least 14 days apart

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women > 18 years of age with a confirmed HIV-1 diagnosis 2. CD4 count <350 and or history of opportunistic infection 3. HIV PCR >55000 and >55,000 on one occasion in last 12 months 4. Patients with poor compliance (Poor compliance will de defined as taking less than 80 percent of prescribed medication 5. Patients with mental illness, HIV dementia, substance abuse or social factor prohibiting compliance 6. Willingness to sign informed consent or legal guardian

-

Exclusion Criteria:

1. ALT/AST > 5X ULN
2. CReatinine >2.0 -

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-04; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Slim, MD, Principal Investigator — Saint Michael's Medical Center
Locations (1):
- Saint Michael's Medical Center, Newark, New Jersey, United States